CLINICAL TRIAL: NCT00168480
Title: A Study Using Botulinum Toxin Type A in Patients With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191622-513
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A

ARMS (1):
- 1 (Experimental): Botulinum Toxin Type A
  Interventions: Biological: Botulinum Toxin Type A

INTERVENTIONS:
Biological: Botulinum Toxin Type A — 100 U, repeated treatments at > 4 month intervals up to Month 32, over a 36-month study period
  Other Names: BOTOX®

SUMMARY:
This is a three year open-label study in subjects with axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Marked axillary hyperhidrosis

Exclusion Criteria:

* Previous use of botulinum toxin for hyperhidrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2003-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Assessment of axillary sweat production | Every 4 Months

SECONDARY OUTCOMES:
Patient reported health outcome measures | 1 Month Post-Treatment Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Portland, Oregon, United States
- Pinneberg, Germany
- Gothenburg, Sweden
- Nottingham, United Kingdom